CLINICAL TRIAL: NCT06207175
Title: A Phase III Trial in Healthy Indonesian Women Ages 18-45 to Evaluate the Immunogenicity and Safety of Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli)
Brief Title: A Study to Evaluate the Immunogenicity and Safety of Nonavalent Human Papillomavirus (HPV) Vaccine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Health Guard Biotechnology, Inc (Industry)
Collaborators: University of Muhammadiyah Malang Hospital (Unknown); Dr. M Djamil Hospital, Padang (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KLWS-V502-05
Record Dates: First submitted 2024-01-02; First posted 2024-01-16 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Human Papillomavirus Infection
Keywords: Human Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections | interventions — Papillomavirus Vaccines; Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The Sponsor, investigators and biostatisticians will remain blinded to subject allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonavalent HPV study vaccine (Experimental): Study vaccine: Recombinant Nonavalent (types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia coli) (Hereinafter referred to as "Nonavalent HPV study vaccine")
  Provided by: Beijing Health Guard Biotechnology, Inc.
  Dosage: 0.5 mL per dose
  Appearance: White, cloudy liquid suspension
  Dosage form: 0.5-mL suspension for injection as a prefilled syringe
  Route of administration: Intramuscular injection into the lateral deltoid muscle of the upper arm
  Vaccination schedule in this study：3 injections on a 0, 2, 6-month schedule.
  Interventions: Biological: Nonavalent HPV study vaccine
- GARDASIL® 9 (Active Comparator): Control vaccine: GARDASIL® 9
  Manufacturer: Merck Sharp and Dohme Corp (MSD).
  Dosage: 0.5 mL per dose
  Appearance: After thorough agitation, GARDASIL® 9 is a white cloudy liquid
  Dosage form: 0.5-mL suspension for injection as a prefilled syringe
  Route of administration: Intramuscular injection into the lateral deltoid muscle of the upper arm
  Vaccination schedule：3 injections on a 0, 2, 6-month schedule.
  Interventions: Biological: GARDASIL® 9

INTERVENTIONS:
Biological: Nonavalent HPV study vaccine — A 3-dose regimen administered at months 0, 2 and 6.
  Other Names: Recombinant Nonavalent (types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia coli)
  Arms: Nonavalent HPV study vaccine
Biological: GARDASIL® 9 — A 3-dose regimen administered at months 0, 2 and 6.
  Arms: GARDASIL® 9

SUMMARY:
This Study to Evaluate the Immunogenicity and Safety of Candidate Recombinant Nonavalent (types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia coli) Administered Intramuscularly in Healthy Female Participants Aged 18 to 45 Years

DETAILED DESCRIPTION:
This is a randomized, observer blinded, active controlled, multicenter clinical study.

A total of approximately 1,260 healthy female participants aged 18 to 45 years old who meet eligibility will be enrolled, and be randomly assigned into 2 groups in a 1:1 ratio.

Immunogenicity: Blood samples (5.0 mL each time) will be collected for all participants prior to the 1st dose of vaccination and on 1, 6, 12, 18 months after full vaccination for anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies and Immunoglobulin G antibodies testing.

Safety evaluation (for all participants):To assess solicited (local and systemic) Adverse Event (AEs) within 7 days after each dose of vaccination, unsolicited Adverse Event (AEs) within 30 days after each dose of vaccination, and Serious Adverse Event (SAEs) from 1st dose to 18 months after full vaccination.

Collection of pregnancy events:To assess the occurrence of pregnancy events in all participants from 1st dose to 18 months after full vaccination. The subject will be followed to determine the outcome of the pregnancy.

At the end of the pregnancy, be it a full-term or premature birth, information on the status of the newborn(s) will be followed up during the first 12 months of life.

ELIGIBILITY:
Inclusion Criteria:

1. *Healthy female participants, aged between 18 years and 45 years as of the 1st dose of vaccination (18 years ≤ age < 46 years).
2. Prior to enrolment, written informed consent obtained from the participants.
3. *Participants must be either of non-childbearing potential, or if of childbearing potential, they must be abstinent or have practiced adequate contraception for 14 days prior to 1st vaccination, and agree to continue such precautions for 1 month after full vaccination.

   [Effective contraception includes oral contraceptives, injectable or implantable contraception, extended-release topical contraceptives, hormonal patches, intrauterine devices (IUDs), sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.]; Women of Childbearing Potential participants have a negative urine pregnancy test before the 1st dose.
4. Participants are able to comply with study protocol, including all scheduled visits, vaccinations, laboratory tests, and other study procedures.

Note: For items with an asterisk (*), If the subject does not meet the criteria, the visit may be rescheduled when the criteria are met.

Exclusion Criteria:

1. * Participant has fever (axillary temperature ≥ 37.3℃) within 24 hours prior to the 1st dose of vaccination;
2. Participant has vaccinated previously or plans to vaccinate with other HPV vaccines during the study period;
3. Participant is participating or plans to participate in other clinical studies during the period of this study;
4. Participant has a history of a positive test for HPV, or a history of an abnormal Pap test result showing atypical squamous cells - undetermined significance (ASC-US), atypical squamous cells - cannot exclude HSIL (ASC-H), low-grade squamous intraepithelial lesion (LSIL), high-grade squamous intraepithelial lesion (HSIL), or atypical glandular cells. Participant has a history of an abnormal cervical biopsy result showing cervical intraepithelial neoplasia (CIN), adenocarcinoma in situ or cervical cancer;
5. Participant has a history of HPV-related genital diseases (e.g., genital warts, Vulvar Intraepithelial Neoplasia, Vaginal Intraepithelial Neoplasia, vulvar cancer, vaginal cancer or anal cancer), a history of venereal disease (e.g., syphilis, gonorrhea, genital chlamydial infection, genital herpes, chancroid, lymphogranuloma venereum, inguinal granuloma, etc.);
6. Participant has a history of allergy to any component of the study vaccine or severe allergic reaction to vaccine (including but not limited to anaphylaxis, allergic laryngeal edema, anaphylactic purpura, thrombocytopenic purpura, or localized allergic necrosis (Arthus reaction), severe urticaria, dyspnea, angioneurotic edema, etc.);
7. Immunocompromised participant or participant that has been diagnosed with congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease, or other autoimmune condition;
8. Participant who has/had epilepsy, excluding a history of febrile seizures under 2 years of age, or alcoholic epilepsy within 3 years prior to alcohol withdrawal;
9. Participant who has severe liver and kidney disease, severe cardiovascular disease, severe diabetes, malignant tumors, severe infectious diseases (e.g., tuberculosis, chronic hepatitis B/C, syphilis, etc.), is unsuitable to participate in this study based on the investigator's judgement;
10. Participant who has thrombocytopenia or any coagulopathy that is not suitable for intramuscular injection;
11. Asplenia or functional asplenia, complete or partial splenectomy from any cause;
12. Participant who is receiving or has received prolonged use (>14 days) of immunosuppressive or other immunomodulatory drugs (e.g., corticosteroids, ≥20 mg/d prednisone or equivalent; however, topical medications such as ointments, eye drops, inhalants or nasal sprays are permitted) within 6 months prior to the 1st dose of vaccination, or plans to receive them during the period from 1st dose of vaccination to 30 days after full vaccination;
13. Participant has received immunoglobulin or other blood products within 3 months prior to the 1st dose of vaccination or plans to receive them during the period from the 1st dose of vaccination to 30 days after full vaccination;
14. *Participant who has acute illness or in acute exacerbation of chronic diseases or use antipyretic, analgesic and anti-allergic drugs (e.g., paracetamol, ibuprofen, aspirin, loratadine, cetirizine, etc.) within 3 days prior to vaccination;
15. *Participant who has vaccinated with inactivated/recombinant/nucleic acid vaccines (non-attenuated vaccines) within 14 days before enrollment or attenuated vaccines within 28 days before enrollment, or plans to administrate vaccine(s) from the 1st dose of vaccination to 30 days after the full vaccination of investigational vaccine.
16. *Participant who donated blood or lost blood ≥ 450 mL within one week before enrollment, or plans to donate blood during the period from the 1st dose of vaccination to 30 days after full vaccination of investigational vaccine;
17. Participant who cannot comply with the requirements of the study due to psychological conditions, and has a history of mental diseases or currently suffer from mental diseases;
18. Participant, who is unsuitable for participation in this study based on the investigator's judgement.

Note: For items with an asterisk (*), if the participant meets these exclusion criteria, the visit may be rescheduled for a time when these criteria are not met. In addition to the examination items set forth in the protocol, other medical history, surgical history and medication history may be obtained in the form of inquiry.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1260 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-11-17 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) for anti-HPV neutralizing antibodies 30 days after full vaccination | 30 days after full vaccination
  Geometric mean titer (GMT) for anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies (pseudo-virus neutralizing assay) 30 days after full vaccination in participants who are seronegative to the relevant HPV type prior to 1st vaccination.
Seroconversion Rate (SCR) for anti-HPV neutralizing antibodies 30 days after full vaccination | 30 days after full vaccination
  Seroconversion Rate (SCR) for anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies (pseudo-virus neutralizing assay) 30 days after full vaccination in participants who are seronegative to the relevant HPV type prior to 1st vaccination.

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of anti-HPV immunoglobulin G antibodies 30 days after full vaccination | 30 days after full vaccination
  Geometric mean titer (GMT) of anti-HPV type 6/11/16/18/31/33/45/52/58 immunoglobulin G antibodies as assessed by enzyme-linked immunosorbent assay (ELISA) 30 days after full vaccination in participants who are seronegative to the relevant HPV type prior to 1st vaccination.
Seroconversion Rate (SCR) of anti-HPV immunoglobulin G antibodies 30 days after full vaccination | 30 days after full vaccination
  Seroconversion Rate (SCR) of anti-HPV type 6/11/16/18/31/33/45/52/58 immunoglobulin G antibodies as assessed by enzyme-linked immunosorbent assay (ELISA) 30 days after full vaccination in participants who are seronegative to the relevant HPV type prior to 1st vaccination.
Geometric mean titer (GMT) of anti-HPV neutralizing antibodies and immunoglobulin G antibodies 6,12,18 months after full vaccination | 6 months, 12 months and 18 months after full vaccination
  Geometric mean titer (GMT) of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies and immunoglobulin G antibodies 6 months, 12 months and 18 months after full vaccination in participants.
Seroconversion Rate (SCR) of anti-HPV neutralizing antibodies and immunoglobulin G antibodies 6,12,18 months after full vaccination | 6 months, 12 months and 18 months after full vaccination
  Seroconversion Rate (SCR) of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies and immunoglobulin G antibodies 6 months, 12 months and 18 months after full vaccination in participants.
Incidenct, severity and duration of each solicited (local and systemic) AE within 7 days after each dose of vaccination | 0-7 days after each dose of vaccination
  Incidenct, severity and duration of each solicited (local and systemic) AE within 7 days after each dose of vaccination.
Incidenct, severity and duration of each unsolicited AE within 30 days after each dose of vaccination | 0-30 days after each dose of vaccination
  Incidenct, severity and duration of each unsolicited AE within 30 days after each dose of vaccination.
Incidence, severity and causality of SAE and incidence of pregnancy events from 1st dose to 18 months after full vaccination | from 1st dose to 18 months after full vaccination
  Incidence, severity and causality of SAE and incidence of pregnancy events from 1st dose to 18 months after full vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hongyang, Study Chair — Beijing Health Guard Biotechnology, Inc
Locations (1):
- University of Muhammadiyah Malang Hospital, Malang, Indonesia

IPD SHARING:
Plan to Share IPD: No
No informed consent was obtained to disclose the subject's data and sample test results